CLINICAL TRIAL: NCT07045675
Title: The Effect of Foot Reflexology Massage on the Perception of Labor Pain in Nulliparous Pregnant Women
Status: Active, not recruiting | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Nurgül Kılıçaslan, mide wife, Atlas University
Other Study IDs: AU-EY-NK-01
Record Dates: First submitted 2025-04-04; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Massage; Labor Pain; Foot Massage; Refleksoloji
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- experimental group: Pregnant women in this group start foot massage when the cervix is 3-4 cm dilated, and this massage is applied 3 times until birth, once when the cervix is 5-8 cm dilated and once when the cervix is 9-10 cm dilated. Massage time for each application is approximately 15 minutes for each foot.
  Pregnant women who agreed to participate in the study were given "Pregnant Introduction Form", "Labor Monitoring Form", "Visual Analogue Scale (VAS)", "Birth Comfort Scale", "State Anxiety Scale", "Postpartum Evaluation Form" and "Birth Satisfaction Scale". "Short Form (DÖ-SHORT FORM)" forms are filled out.
- control group: Massage is not applied to pregnant women in this group. Only forms are filled out.
  Pregnant women who agreed to participate in the study were given "Pregnant Introduction Form", "Labor Monitoring Form", "Visual Analogue Scale (VAS)", "Birth Comfort Scale", "State Anxiety Scale", "Postpartum Evaluation Form" and "Birth Satisfaction Scale". "Short Form (DÖ-SHORT FORM)" forms are filled out.

SUMMARY:
To evaluate the effect of reflexology massage, which is a non-pharmacological tool based on the effect of reflexology massage applied to the foot, on the perception of labor pain, on the perception of labor pain.

DETAILED DESCRIPTION:
This research; It was planned as an experimental prospective randomized controlled clinical study to determine the effect of reflexology massage applied with the relaxation technique in the first stage of labor on perceived labor pain.

hypotheses H₁; There is a difference in perceived labor pain between the experimental group that received reflexology massage during labor and the control group.

H₂; There is a difference in birth times between the experimental group and the control group, which received reflexology massage during labor.

H₃; There is a difference in the level of state anxiety between the experimental group and the control group, which received reflexology massage during labor.

H₄; There is a difference in the level of postpartum fatigue between the experimental group and the control group, which received reflexology massage during labor.

H₅; There is a difference in the level of birth satisfaction between the experimental group and the control group, which received reflexology massage during labor.

H₆; There is a difference between the experimental group, which received reflexology massage during labor, and the control group, in terms of the time it takes to initiate breastfeeding in the postpartum period.

H₇; There is a difference in comfort levels at birth between the experimental group and the control group, which received reflexology massage during labor.

ELIGIBILITY:
Inclusion Criteria:Pregnancy at term (37-42 weeks)

* Having a single, live fetus in vertex position
* Being in the latent phase of labor
* Cervical dilation is less than 5 cm
* Planning vaginal birth
* No pregnancy complications
* Contractions have started and are regular
* No language problems
* Able to communicate verbally
* Pregnant women who agree to work.

Exclusion Criteria:

Narcotic analgesic or sedative area

* Those with systemic diseases such as heart disease, hypertension, diabetes, kidney disease
* Pregnant women with pregnancy complications (placenta previa, preeclampsia, oligohydramnios, polyhydramnios, position/presentation disorder, etc.).

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — nulliparous pregnant women
Study Population: 717
Sampling Method: Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
Vizüel Analog Skala (VAS) | from the 1st stage of labor to birth
  The most common VAS consists of a 10 cm horizontal or vertical line with two ends labeled "no pain" and "worst possible pain" (or similar verbal descriptors). Patients are asked to place a mark on a point on a 10 cm line that corresponds to the level of pain intensity they feel. The distance in centimeters from the lower end of the VAS to the mark placed by the patient is used as the numerical value of pain intensity.
Pregnant Introduction Form | from the 1st stage of labor to the 2nd hour after birth
  By scanning the literature, there are a total of 39 questions: 10 questions covering the sociodemographic characteristics of the pregnant woman, 17 questions covering her medical and obstetric characteristics, and 12 questions covering her knowledge and thoughts about birth.
Labor Follow-up Form | from the 1st stage of labor to the 2nd hour after birth
  In the labor follow-up form; week of gestation, date and time when labor pains started, medications and applications administered in the first stage of labor, table of evaluations before and after reflexology massage application (cervical dilatation and effacement, head level and condition of membranes, intensity and frequency of contractions, fetal heart rate ( FKA), the mother's vital signs and behaviors during labor), the start time of the 2nd stage, the end time, the total duration of labor, questions regarding the first evaluation of the newborn (baby's gender, head circumference, weight, height, APGAR score and health status, initiation of the first breastfeeding and the mother's breastfeeding status).
Birth Comfort Scale | from the 1st stage of labor to the 2nd hour after birth
  It consists of questions about pregnant women's opinions about their birth comfort during VM. The Cronbach Alpha coefficient of the scale was found to be 0.75. 24 The Cronbach Alpha coefficient of this study was found to be 0.72. The scale consists of 9 questions and is in the 5-point Likert type (1 = Totally disagree, 2 = Mostly disagree, 3 = Partially agree, 4 = Mostly agree, 5 = Completely agree). It is expected that the items will be answered considering the comfort in the delivery room. Each expression communicates a specific feeling of comfort (relaxation, relief, or superiority) and dimensions (physical, environmental, psychospiritual, or social). A minimum of 9 and a maximum of 45 points are obtained from the scale. It is stated that as the
Postpartum Evaluation Form | from the 1st stage of labor to the 2nd hour after birth
  Postpartum evaluation form; It was prepared to evaluate the birth process for participants in the DSO group and control group. It is administered at the 2nd hour after birth and includes questions about the pregnant woman's thoughts about this birth, her thoughts about labor pain, how they feel after birth, and their satisfaction with the practices performed during labor.
Birth Satisfaction Scale Short Form | from the 1st stage of labor to the 2nd hour after birth
  The Short Form of the Childbirth Satisfaction Scale is a 10-question, 5-point Likert-type scale, consisting of 3 sub-dimensions: "quality of care", "stress during labor" and "personal characteristics of the woman". The "quality of care services" sub-dimension is measured with items 3, 5, 6 and 10, the "stress during labor" sub-dimension with items 1, 2, 7 and 9, and the "personal characteristics of the woman" sub-dimension with items 4 and 8. It is scored as "strongly disagree" (0 points), "disagree" (1 point), "undecided" (2 points), "agree" (3 points), and "strongly agree" (4 points). Scores range from 0 to 40 on the scale, and as the score increases, the satisfaction level increases; low satisfaction <13 points, medium satisfaction 14-27 points, and high satisfaction ≥28 points. 6 items in the scale are positive, 4 items are negative, and 4 items (2nd, 4th, 7th, 8th) are scored in reverse. The Cronbach alpha level of the scale was found to be 0.682.

CONTACTS AND LOCATIONS:
Overall Officials: nurgül kılıçaslan, Principal Investigator — İstanbul Kanuni Sultan Süleyman Eğitim ve Araştırma Hastanesi
Locations (1):
- İstanbul Kanuni Sultan Süleyman Eğitim ve Araştırma Hastanesi, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The decision will be made according to the study results.

REFERENCES:
- See also: Related Info — https://dergipark.org.tr/tr/pub/akd/issue/67025/1047261#article_cite